CLINICAL TRIAL: NCT05684237
Title: Using the VisuMax Femtosecond Laser System to Perform SMILE Optimized for Presbyopia by Modulation of Postoperative Spherical Aberration
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: London Vision Clinic (Other)
Responsible Party: Principal Investigator, Dan Reinstein, Medical Director, London Vision Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LoVC-010
Record Dates: First submitted 2022-12-21; First posted 2023-01-13 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Myopia; Myopic Astigmatism; Presbyopia
MeSH Terms: conditions — Myopia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HiSMILE treatment option (Other): HiSMILE treatment option
  Interventions: Procedure: HiSMILE treatment option

INTERVENTIONS:
Procedure: HiSMILE treatment option — The non-CE labeled VisuMax treatment option HiSMILE is able to modify the lenticule shape in a way that should lead to a change in spherical aberration postoperatively.

SUMMARY:
The intended purpose of the investigational device in the study is the correction of myopia and myopia with astigmatism in the CE (Conformité Européene) approved range and optimized for presbyopic patients using the treatment option HiSMILE, installed on the VisuMax femtosecond laser.

DETAILED DESCRIPTION:
Presbyopia refers to an impairment of near vision that is common among adults over 40 years of age. It is known to considerably decrease quality of life, especially given the heavy use of computers and smartphones. The management of presbyopia can be divided into non-surgical approaches, such as glasses and contact lenses, and surgical approaches.

A refractive surgical approach to treating presbyopia was developed by Reinstein et al termed PRESBYOND® Laser Blended Vision. PRESBYOND® is different from traditional monovision (when the dominant eye is mainly corrected for distance and the non-dominant eye is mainly corrected for near) because it increases the depth of field as a result, a blend zone is created, which allows the patient to see near, intermediate and far without glasses

Following its introduction in 2011, surgical approaches such as small incision lenticule extraction (SMILE) are increasing in popularity due to the high level of safety, efficacy and other advantages. Compared to laser-assisted in situ keratomileusis (LASIK), SMILE preserves more corneal nerves and better maintains the strength of the cornea. Worldwide more than 6 million SMILE procedures have been performed.

SMILE has also been combined with monovision as a treatment option for presbyopic patients. First results of SMILE monovision in patients with presbyopia and short-sightedness (myopia) have been published showing promising outcomes for distance and near vision. However, those investigations noted SMILE did not increase the depth of field, and as a result outcomes for vision at the intermediate (computer) distance did not reach the level as those achieved with PRESBYOND LASIK.

Therefore, a new treatment option called HiSMILE was developed to improve the depth of field and therefore the intermediate vision. A clinical study is required to investigate whether the HiSMILE treatment option can alter the depth of field for different levels of short-sightedness to achieve the required levels without compromise to contrast sensitivity or quality of vision.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfillment of the general inclusion criteria stated in User Manual of the VisuMax option SMILE
2. Presence of myopia up to -10.00 D with or without astigmatism up to 5.00 D and a maximum spherical equivalent of -12.50 D (SMILE CE approved range)
3. Age of 40 years or older
4. Presence of presbyopia
5. Patients able to receive a refractive correction in both eyes and in addition a compensation of presbyopia, in which one eye should be targeted for far vision and one eye should be targeted for near vision
6. Pre-operative CDVA of 20/25 or better in each eye as well as a Distance Corrected Near Visual Acuity (DCNVA) of 20/25 (J2) or worse
7. Target refraction of the near eye between -0.50 D to -1.75 D
8. Acceptance of anisometropia (no visual discomfort or disturbances during the Acceptance Test before surgery, eye intended for near vision determined during this test)
9. Compliance with follow-up visits and examinations

Exclusion Criteria:

1. Presence of at least one of the contraindications stated in the User Manual of the VisuMax option SMILE or in the Surgical Information Package provided to the patient by the London Vision Clinic before surgery
2. Hyperopic refraction
3. Mixed astigmatism refraction
4. Emmetropic eyes, defined as spherical equivalent refraction <-0.88 D, maximum hyperopia ≤+1.00 D and cylinder <1.25 D
5. Patients presenting any kind of amblyopia
6. Previous intraocular or corneal surgery
7. Participation in other ophthalmologic or pharmaceutical studies
8. Women during pregnancy and/or lactation
9. Patients whose freedom is impaired by administrative or legal order
10. Persons incapable of giving consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Performance | 3 Months
  Percentage of eyes with ocular spherical aberration within the therapeutic range of 0.3 to 0.6 μm (Optical Society of America notation at 6 mm analysis diameter) at 3 months.
Performance | 12 Months
  Percentage of eyes with ocular spherical aberration within the therapeutic range of 0.3 to 0.6 μm (Optical Society of America notation at 6 mm analysis diameter) at 12 months.
Safety Outcome | 3 Months
  Percentage of eyes with loss of 2 lines (10 letters) or more of Corrected Distance Visual Acuity (CDVA) at 3 months postoperative compared to the baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Dan Reinstein, Principal Investigator — London Vision Clinic
Locations (1):
- London Vision Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No